CLINICAL TRIAL: NCT02175628
Title: Comparison of the Sensitivity and Specificity of Acoustic Angiography (Micro-tumor Detection by Quantifying Tumor-induced Vascular Abnormalities) to the Sensitivity and Specificity of Conventional Ultrasound
Brief Title: Comparison of the Sensitivity and Specificity of Acoustic Angiography to the Sensitivity and Specificity of Conventional Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1405; R01CA170665 (NIH)
Record Dates: First submitted 2014-06-20; First posted 2014-06-26 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2018-10

CONDITIONS: Signs and Symptoms
Keywords: Ultrasound; Breast; Angiography
MeSH Terms: conditions — Signs and Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acoustic Angiography (Experimental): All breast patients will be included in the experimental group.
  Interventions: Device: Acoustic Angiography
- Healthy Volunteers (Experimental): A volunteer group was added to the study to perfect the image acquisition techniques.
  Interventions: Device: Acoustic Angiography

INTERVENTIONS:
Device: Acoustic Angiography — Acoustic angiography imaging involves a research high frequency ultrasound scanner (VisualSonics Vevo 770) and a prototype transducer as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. The imaging also requires administration of Definity ultrasound contrast agent.
  Acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion. Total imaging time is estimated to be less than 15 minutes. All image data will be de-identified and transferred for off-line analysis based on a study ID. The research images will NOT be interpreted or analyzed for clinical decisions related to the patient.

SUMMARY:
Purpose: This study will evaluate a new ultrasound imaging technology called acoustic angiography. Acoustic angiography uses an ultrasound contrast agent, already FDA approved for use in cardiology, to enhance imaging of blood vessels. Since acoustic angiography uses ultrasound, and not x-rays, the patient is not exposed to ionizing radiation, unlike traditional angiography and mammography. Specific goals will be to evaluate the quality of the images provided by acoustic angiography in the human breast, and furthermore to evaluate whether or not acoustic angiography provides additional diagnostic information over traditional ultrasound which could provide an improvement in assessing breast lesions. Specifically, this additional diagnostic information will hopefully enable us to reduce false positive tests and discriminate lethal cancers from non-lethal disease.

Participants: The investigators are recruiting 60 patients from the UNC Breast Clinic who are undergoing core needle biopsy or surgical biopsy (BIRADS 4 and 5 breast lesions).

Procedures (methods): Acoustic Angiography imaging will be performed in conjunction with standard diagnostic imaging, including b-mode ultrasound . Then, a reader study will be conducted to compare these modalities. Finally, the images will be analyzed with image processing techniques to determine quantitative metrics exhibited by the blood vessel morphology in the images. These metrics will be utilized to develop a "malignancy score" equation to predict malignancy of a lesion.

DETAILED DESCRIPTION:
Increasing the sensitivity and specificity of diagnostic imaging in patients at high risk for breast cancer could provide substantial clinical benefit by improving diagnosis, preventing over-treatment, and reducing healthcare costs. Acoustic angiography is a new type of contrast enhanced ultrasound imaging which is specifically sensitive to microvascular structure and density. It evaluates tumor micro-vasculature and may provide a powerful prognostic tool for the diagnosis of breast cancer, and eventually for treatment evaluation.

Sixty patients who are to have a clinical surgical breast biopsy based on results from pre-study standard of care (SOC) imaging will be recruited from the UNC Breast Clinic for participation in the study. The primary objective of this single arm study is to compare the sensitivity and specificity of acoustic angiography with traditional b-mode ultrasound in the distinction of malignant versus benign breast lesions. Secondary objectives include a comparison of area under the curve (AUC) for acoustic angiography versus b-mode ultrasound, comparison of radiologist preference for the two imaging techniques for each of 3 lesion characteristics, and quantification of vessel tortuosity based on acoustic angiography imaging results. These metrics will be used to develop a predictive model of malignancy which will subsequently be compared to results from radiology review.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years old
* Scheduled for breast core needle or surgical biopsy of at least one breast lesion based on suspicious breast lesion (BIRADS score of 4 or 5) from pre-study SOC imaging studies
* Center of suspicious lesion is not deeper than 1.5 cm, and the diameter of the lesion is not greater than 2 cm
* Able to provide informed consent
* Negative urine pregnancy test in women of child-bearing potential

Exclusion Criteria:

* Male (it is uncommon for men to present for imaging and the overwhelming majority of findings are non-cancerous and do not lead to biopsy; male breast cancer represents <1% of newly diagnosed breast cancer)
* Institutionalized subject (prisoner or nursing home patient)
* Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD)
* Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®)
* Right to left shunt, severe pulmonary hypertension (pulmonary artery pressure >90mmHg), or adult respiratory distress syndrome
* Active cardiac disease including any of the following:

  * Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
  * Unstable angina.
  * Severe arrhythmia (i.e. ventricular tachycardia, flutter fibrillation; ventricular premature complexes occurring close to the preceding T-wave, multifocal complexes).
  * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
  * Uncontrolled systemic hypertension (systolic blood pressure (BP) >150 mm Hg and/or diastolic BP >90 mm Hg despite optimal medical management

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Lee, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospital, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acoustic Angiography: All breast patients will be included in the experimental group.
  Acoustic Angiography: Acoustic angiography imaging involves a research high frequency ultrasound scanner (VisualSonics Vevo 770) and a prototype transducer as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. The imaging also requires administration of Definity ultrasound contrast agent.
  Acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion. Total imaging time is estimated to be less than 15 minutes. All image data will be de-identified and transferred for off-line analysis based on a study ID. The research images will NOT be interpreted or analyzed for clinical decisions related to the patient.
- Healthy Volunteers: A volunteer group was added to the study to perfect the image acquisition techniques.
  Acoustic Angiography: Acoustic angiography imaging involves a research high frequency ultrasound scanner (VisualSonics Vevo 770) and a prototype transducer as well as conventional b-mode ultrasound to guide the location of the imaging. The conventional ultrasound will be conducted just prior to the acoustic angiography for localization. The imaging also requires administration of Definity ultrasound contrast agent.
  Acoustic angiography imaging will be performed by trained medical personnel using mild compression to eliminate motion. Total imaging time is estimated to be less than 15 minutes. All image data will be de-identified and transferred for off-line analysis based on a study ID. The research images will NOT be interpreted or analyzed for clinical decisions related to the patient.
Period: Overall Study
Arm/Group | Acoustic Angiography | Healthy Volunteers
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acoustic Angiography | Healthy Volunteers | Total
Number analyzed (Participants) | 6 | 17 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 15 | 20
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (14) | 43 (17) | 45 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 8 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 10 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 17 | 23

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity (Percentage)
Description: To compare (using a reader study) the sensitivity and specificity of acoustic angiography to the sensitivity and specificity of conventional b-mode ultrasound in evaluation of breast lesions
Time Frame: 1.5 years
Population: The data were unable to be analyzed because we could not visualize the vessels to calculate this value. The system was unable to achieve the imaging resolution to visualize the vasculature.
Arm/Group | Acoustic Angiography | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Area Under the Curve (AUC) of Acoustic Angiography
Description: The AUC of acoustic angiography compared to the AUC of b-mode ultrasound
Time Frame: 1.5 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Radiologist Preference
Description: To compare radiologist preference of acoustic angiography to conventional b-mode ultrasound for each lesion characteristic (shape, margins and vascularity)
Time Frame: 1.5 years
Population: Preference Study not conducted because the imaging resolution was insufficient. The data were unable to be analyzed because we could not visualize the vessels to calculate this value. The system was unable to achieve the imaging resolution to visualize the vasculature.
Arm/Group | Acoustic Angiography | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vessel Tortuosity (No Units)
Description: To quantify vessel tortuosity metrics for the acoustic angiograph images, and to use these metrics to develop a model for predicting malignancy (a model-based malignancy score)
Time Frame: 1.5 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Model-based Malignancy Score (Arbitrary Units)
Description: To compare the model-based malignancy score to the acoustic angiography reader study
Time Frame: 1.5 years
Population: as for outcome 1
Arm/Group | Acoustic Angiography | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 minutes post imaging
Arm/Group | Acoustic Angiography | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/17
Other Adverse Events (participants affected / at risk) | 0/6 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT02175628/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02175628/ICF_001.pdf